CLINICAL TRIAL: NCT07020520
Title: EvaluatioN of Optilume Drug-Coated Balloon for the Endoscopic Treatment of UREteric Strictures
Acronym: ENDURE1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Urotronic Inc. (Industry)
Collaborators: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1391
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Ureteral Stricture
Keywords: ureteral; ureteric; stricture; stenosis; optilume
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: There is a main study and pharmacokinetic (PK) substudy. All subjects will receive the same treatment. PK substudy subjects (15) will also have serum and urine samples collected for analysis of paclitaxel levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Optilume (Experimental): Treatment with Optilume for ureteric stricture
  Interventions: Device: Optilume

INTERVENTIONS:
Device: Optilume — Has pre-treatment (balloon dilation or ureterotomy) followed by paclitaxel-coated balloon (Optilume) treatment of the ureteric stricture.

SUMMARY:
The main objective of this clinical investigation is to assess the safety and feasibility of the Optilume DCB for treatment of ureteric strictures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Single lesion ureteric or uretero-enteric stricture less than or equal to 4.0 cm in length
3. Two functioning kidneys

Exclusion Criteria:

1. Treatment of the target ureter with incision or balloon dilation within 3 months of the study treatment
2. Subjects with more than one ureteric stricture
3. Subjects with target stricture in bifid or duplicated ureter
4. Known sensitivity to paclitaxel or on medication that may have negative interaction with paclitaxel
5. Ureteric stricture caused by extrinsic compression of the ureter
6. Unable to endoscopically access target stricture for any reason
7. Existing stones in the ipsilateral kidney or ureter (except for asymptomatic kidney stones) that are in close proximity to the target ureteric stricture
8. Chronic renal failure treated with dialysis
9. eGFR <30 mL/min/1.73m2
10. Kidney function ≤ 25% of split function on the side with target stricture as measured by functional renogram
11. Kidney function ≤35% of split function on the side opposite target stricture as measured by functional renogram or other significant pathology or impairment that may impact renal function
12. Life expectancy less than 12 months
13. Women who are pregnant or breastfeeding
14. Women of child-bearing potential planning to get pregnant in the next year or are unwilling to use contraception over the next 12 months
15. Males unwilling to abstain or use protected sex for 30 days post treatment
16. Males unwilling to use highly effective contraception for6 months post treatment if sexual partner(s) are of child-bearing potential
17. Inability to provide legally effective informed consent
18. Unwilling or unable to meet protocol follow-up requirements
19. Participation in any interventional clinical investigation of a medical device, drug, or biologic (excluding registries) that may confound the results of the trial
20. Active systemic or urinary tract infection
21. Active malignancy in the abdomen or pelvis, or any malignancy considered considerable risk for metastasizing to the abdomen or pelvis over the next 12 months
22. Uncontrolled diabetes defined as hemoglobin A1C ≥ 8% at baseline
23. Unable to come off antiplatelet or anticoagulation medication prior to treatment to prevent bleeding complications at the discretion of the investigator
24. Any other condition that may confound the results of the trial or presents an unacceptable risk for any study-related procedure
25. Individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response
26. Presence of any condition that precludes administration of furosemide during renograms
27. Unable to tolerate contrast related to required study procedures or imaging.

Additional Criteria for Pharmacokinetic Substudy Inclusion Ureteric stricture measurements appropriate for treatment with a 6mm (18F) or 8mm (24F) diameter Optilume DCB Exclusion Prior treatment with any device or medical therapy that contains paclitaxel, including drug coated balloons for vascular and urethral applications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
Successful treatment | 6-months post ureteral stent removal (approximately 7 months post Optilume treatment)
  Rate of successful treatment defined as meeting all the following criteria:
  * Technical success
  * Freedom from retreatment of target stricture through six months post stent removal
  * Renogram at 6 months showing stability or improvement in split function for impacted kidney defined as split function within 10% of baseline value or improved from baseline.
  * T1/2 stability or improvement from baseline to 6 months for impacted kidney

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Landman, MD, Principal Investigator — University of California, Irvine
Locations (5):
- United States (5):
  - University of California Irvine, Orange, California
  - Orlando Health, Orlando, Florida
  - Mount Sinai, New York, New York
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No